CLINICAL TRIAL: NCT04676425
Title: A 2-part, Open-label, Single-dose Study to Investigate the Influence of Hepatic Impairment on the Pharmacokinetics of MK-8189
Brief Title: A Study to Investigate the Influence of Hepatic Impairment on MK-8189 Treatment (MK-8189-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8189-012; MK-8189-012 (Other: Merck)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-12

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — MK-8189

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Hepatic Impairment Participants (Experimental): Participants with hepatic impairment will receive a single dose of MK-8189 4 mg orally on Day 1.
  Interventions: Drug: MK-8189
- Healthy Participants (Experimental): Healthy participants will receive a single dose of MK-8189 4 mg orally on Day 1.
  Interventions: Drug: MK-8189

INTERVENTIONS:
Drug: MK-8189 — Administered at a dose of 4 mg via oral tablet

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (PK) of MK-8189 in participants with moderate hepatic impairment (based on the Child-Pugh classification) to healthy participants. This is Part 1 of the study; following review of the safety and PK data from Part 1, a decision will be made as to whether Part 2 of the study will be initiated. If done, Part 2 of the study will compare the PK of MK-8189 in participants with mild hepatic impairment to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Is a continuous non-smoker or moderate smoker (of fewer than 20 cigarettes/day or equivalent)
* Female participant is not pregnant or breastfeeding and is not woman of childbearing potential (WOCBP) or is a WOCBP using contraception or abstinent from heterosexual intercourse during the intervention period and for at least 14 days after the last dose of study intervention
* (For hepatically impaired participants) Has a diagnosis of chronic (>6 months), stable (no acute episodes within the previous 2 months due to deterioration in hepatic function) hepatic impairment

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormalities or diseases
* Has a history of cancer; exceptions include (1) adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix, (2) other successfully treated malignancies
* Has a history of significant multiple and/or severe allergies or has had significant intolerability to prescription or non-prescription drugs or food
* Is positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Has had major surgery or lost 1 unit of blood within 4 weeks prior to prestudy visit
* Consumes greater than 3 glasses of alcoholic beverages per day
* Consumes greater than 6 servings (1 serving is ~120 mg of caffeine) caffeinated beverages per day
* (For hepatically impaired participants) Is taking medications to treat chronic medical conditions and has not been on a stable regimen for at least 1 month and/or is unable to withhold the use of the medications during study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - ProSciento Inc. ( Site 0002), Chula Vista, California
  - Clinical Pharmacology of Miami ( Site 0001), Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As prespecified in the protocol, the safety and pharmacokinetic (PK) data from Part 1 of the study, comparing participants with moderate hepatic impairment to healthy participants, were reviewed after completion of Part 1. Per protocol, a decision was made to not conduct Part 2 of the study, comparing participants with mild hepatic impairment to healthy participants.
Groups:
- Moderate Hepatic Impairment Participants: Participants with moderate hepatic impairment received a single dose of MK-8189 4 mg orally on Day 1.
- Healthy Participants: Healthy participants received a single dose of MK-8189 4 mg orally on Day 1.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (8.2) | 57.1 (8.0) | 56.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MK-8189
Description: AUC0-inf is a measure of the total amount of drug in the plasma from the dose administration extrapolated to infinity. Blood samples collected pre and post-dose at multiple timepoints were used to estimate AUC0-inf following MK-8189 administration. Geometric least-squares mean and confidence intervals for AUC0-inf were calculated using a linear fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose (0), 2, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose (hepatic impairment and healthy participants); 60, 84, 108 and 120 hours post-dose (hepatic impairment participants)
Population: All participants who were compliant with the study procedures and have available data from at least one treatment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*nmol/L
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants
Number analyzed (Participants) | 7 | 7
h*nmol/L | 5600 [3020 to 10400] | 4710 [3340 to 6660]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Participants vs Healthy Participants; Test type: Other; Least-Squares Geometric Mean Ratio = 1.19, 90% CI 2-sided [0.70 to 2.01] — Moderate hepatic impairment participants represent the numerator and healthy participants represent the denominator in the geometric mean ratio

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of MK-8189
Description: Cmax is the maximum concentration of MK-8189 observed in plasma. Blood samples collected pre and post-dose at multiple timepoints were used to estimate Cmax following MK-8189 administration. Geometric least-squares mean and confidence intervals of Cmax were calculated using a linear fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose (0), 2, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose (hepatic impairment and healthy); 60, 84, 108 and 120 hours post-dose (hepatic impairment)
Population: All participants who were compliant with the study procedures and have available data from at least one treatment
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants
Number analyzed (Participants) | 7 | 7
nmol/L | 194 [127 to 296] | 158 [131 to 191]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Participants vs Healthy Participants; Test type: Other; Least-Squares Geometric Mean Ratio = 1.22, 90% CI 2-sided [0.86 to 1.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs will be reported.
Time Frame: Up to approximately 15 days
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants
Number analyzed (Participants) | 7 | 7
Participants | 4 | 0

4. Secondary Outcome: Number of Participants Who Discontinue From the Study Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study due to an AE will be reported.
Time Frame: Up to approximately 15 days
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 15 days
Description: All participants who received at least one dose of treatment are included
Arm/Group | Moderate Hepatic Impairment Participants | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment Participants (N=7) | Healthy Participants (N=7)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT04676425/Prot_SAP_000.pdf